CLINICAL TRIAL: NCT00123695
Title: Serial Echocardiography After Subarachnoid Hemorrhage (S.E.A.S.)
Brief Title: Serial Echocardiography After Subarachnoid Hemorrhage
Acronym: SEAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other)
Other Study IDs: 04-193
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Subarachnoid Hemorrhage; Myocardial Stunning; Takotsubo Cardiomyopathy
Keywords: Subarachnoid hemorrhage; Takotsubo cardiomyopathy; Cardiac abnormalities; outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage; Myocardial Stunning; Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is increasing interest in myocardial abnormalities following central nervous system events, such as subarachnoid hemorrhage (SAH). These cardiac abnormalities include ECG changes, decreased cardiac output, decreased blood pressure, specific cardiac enzyme elevations, and segmental wall motion abnormalities (SWMA). Interestingly, wall motion abnormalities and ECG changes have shown to be reversible, and therefore the dysfunction has been described as neurogenic myocardial stunning.

The pathophysiology of cardiac dysfunction following SAH has not yet been fully elucidated. Many reports (mainly case reports) have been published, but so far no study has investigated the frequency of these abnormalities in a prospective manner, have correlated the occurrence of the different cardiac abnormalities, and have assessed which clinical variables can predict cardiac dysfunction. And only a limited number of studies have related neurological outcome with cardiac dysfunction.

DETAILED DESCRIPTION:
Objectives: Therefore, our study objectives are: 1) Assessment of the frequency of myocardial dysfunction (segmental wall motion abnormalities, cardiac-specific enzyme elevations, and ECG changes) in patients with SAH. 2) Determination of predictive clinical variables for the occurrence of myocardial dysfunction following SAH. 3) Impact of myocardial dysfunction on neurological prognosis: death, secondary cerebral ischemia, hydrocephalus and rebleeding.

Methods: For this purpose serial echocardiograms and ECGs will be obtained and cardiac enzymes will be measured in 200-400 patients admitted to hospital with SAH in the four participating centers. The clinical variables that will be studied to predict cardiac dysfunction are: medical history, the CT-scan score, circulatory parameters, blood samples, medication, surgical intervention (coiling or clipping), and the neurological condition (Glasgow Coma Scale). The echocardiograms, ECGs and cardiac enzymes will be studied to determine if they have independent prognostic value for the outcome in SAH patients.

Expected Results: As ECG changes and drops in blood pressure are known to occur frequently, the researchers expect to find that cardiac contractile dysfunction in patients with SAH occurs more frequently than is assumed now. Moreover, if cardiac abnormalities have neurological prognostic significance further studies are needed for early recognition and treatment of the cardiac abnormalities in SAH, a condition with a very poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with aneurysmal subarachnoid hemorrhage
* Admitted within 72 hours of the bleed

Exclusion Criteria:

* No informed consent
* Patients or patients' family unwillingness to participate

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frans C Visser, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc; Ivo A van der Bilt, MD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Gabriel J Rinkel, MD PhD, Principal Investigator — UMC Utrecht; Arthur A Wilde, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (6):
- Netherlands (6):
  - Academic Medical Center, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center Rotterdam, Rotterdam
  - Saint Elisabeth Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] van der Bilt IA, Hasan D, van den Brink RB, Cramer MJ, van der Jagt M, van Kooten F, Regtien JG, van den Berg MP, Groen RJ, Cate FJ, Kamp O, Gotte MJ, Horn J, Girbes AR, Vandertop WP, Algra A, Rinkel GJ, Wilde AA; SEASAH (Serial Echocardiography After Subarachnoid Hemorrhage) Investigators. Time course and risk factors for myocardial dysfunction after aneurysmal subarachnoid hemorrhage. Neurosurgery. 2015 Jun;76(6):700-5; discussion 705-6. doi: 10.1227/NEU.0000000000000699. PMID 25714519